CLINICAL TRIAL: NCT06643260
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Efficacy and Safety of Daily Piclidenoson (CF101) Administered Orally in Subjects With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Phase 3 Study in Moderate-to-Severe Plaque Psoriasis With Piclidenoson to Study Safety and Efficacy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-302PS
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Plaque Psoriasis
Keywords: Psoriasis; Plaque psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: This trial will be conducted in 2 sequential Segments. When the planned number of subjects have completed Segment 1, enrollment will be paused to perform an interim analysis for futility. If futility is not declared, enrollment in Segment 2 will commence. There will be one decision made in this futility analysis that will be conducted by an outside committee. Blinding will remain in full except for a select group of this committee. The committee will decide either to stop the study because of futility, continue the study as is, or continue the study with an increase in sample size. The increase in sample size cannot be greater than 25% of the planned sample size.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Piclidenoson treatment (Experimental)
  Interventions: Drug: piclidenoson
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: piclidenoson — Piclidenoson is a selective A3AR agonist, supplied as tablets.
  Arms: Piclidenoson treatment
Drug: Placebo — Inactive control
  Arms: Placebo

SUMMARY:
This is a double-blind, placebo-controlled study in adults with a diagnosis of moderate-to-severe chronic plaque psoriasis to test the efficacy and safety of piclidenoson in this patient population.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study in adult males and females, aged 18 years and above, with a diagnosis of moderate-to-severe chronic plaque psoriasis.

This trial will be conducted in 2 sequential Segments. When the required number of subjects have completed Segment 1, enrollment will be paused to perform an interim analysis for futility. If futility is not declared, enrollment in Segment 2 will commence. No subject will participate in both Segment 1 and Segment 2.

For subjects in Segment 1, the design is as follows:

At the Screening Visit (Visit 1, performed within 4 weeks prior to randomization), subjects who provide written informed consent will have screening procedures performed, including a complete medical history, medication history, physical examination (including height, weight, sitting blood pressure, respiratory rate, pulse rate and temperature), ECG, Patient Health Questionnaire-9 (PHQ-9), Columbia Suicide Severity Rating Scale (C-SSRS), and assessment of psoriasis (including Psoriasis Area and Severity Index (PASI), Static Physician's Global Assessment (sPGA), Body Surface Area (BSA) involved, Psoriasis Symptoms and Signs Diary (PSSD), and Dermatology Life Quality Index (DLQI)), and clinical laboratory tests.

For subjects enrolled in Segment 2, the design is as follows:

At the Screening Visit (Visit 1, performed within 4 weeks prior to randomization), subjects who provide written informed consent will have screening procedures performed, including a complete medical history, medication history, physical examination (including height, weight, sitting blood pressure, respiratory rate, pulse rate and temperature), ECG, PHQ-9, C-SSRS, and assessment of psoriasis [including PASI score, sPGA, BSA involved, PSSD, DLQI, Psoriasis Scalp Severity Index (PSSI) (for subjects with scalp involvement), and Nail Psoriasis Severity Index (NAPSI) (for subjects with nail involvement)], and clinical laboratory tests.

The trial for Segment 2 subjects will be conducted in 3 Periods: Period A (Primary Efficacy Period, Weeks 0-16), Period B (Crossover Period, Weeks 17-32), and Period C (Randomized Withdrawal Period, Weeks 33-52).

For the patients included in Segment 1 of the trial, only Period A (Primary Efficacy Period, Weeks 0-16) will be applicable.

For the patients included in Segment 2 of the trial, all the 3 study periods A, B and C will be applicable.

In Period A (both Segments), subjects will be randomized in a 2:1 ratio (active:placebo) to receive oral piclidenoson 3 mg or matching placebo twice a day (BID) in double-blinded fashion. The primary efficacy evaluation will occur at the end of Period A/Week 16 visit.

In Period B (Segment 2 only), beginning at the Week 16 visit, all subjects initially assigned to the placebo group will be switched to piclidenoson 3 mg BID.

At the Week 24 visit and beyond (including Period C), subjects who do not achieve and maintain at least a PASI 50 response will be withdrawn from dosing.

In Period C (Segment 2 only), subjects who were initially randomized to piclidenoson and achieve PASI 75 (a ≥75% reduction from Baseline in PASI) OR an sPGA of 0 or 1 with at least a 2-point improvement from Baseline at Week 32 will be rerandomized (1:1, blinded) to continue piclidenoson or switch to placebo (i.e., treatment withdrawal). Subjects rerandomized to placebo at Week 32 will resume piclidenoson if, at any in-clinic visit before Week 52, they lose treatment response, defined as losing at least 50% of the PASI improvement (absolute numerical score) experienced at Week 32 compared to Baseline PASI score; OR an sPGA ˃ 1. Subjects who were initially randomized to placebo in Period A and crossed over to piclidenoson in Period B will continue piclidenoson through Period C (i.e., through Week 52).

At Week 32 and every in-clinic visit thereafter, subjects with less than PASI 75 response (PASI <75) or an sPGA ˃ 1, regardless of initial treatment or current study drug treatment, will be allowed to add topical treatment such as salicylic acid and low-potency or weak corticosteroids (US Class 6 or 7, such as hydrocortisone, desonide, alclometasone dipropionate) and/or ultraviolet B phototherapy, per Investigator judgment.

Blinding for Period A (Primary Efficacy Period) will be maintained for the duration of the trial, defined as all subjects (Segment 1 and Segment 2) having completed all of their visits. Due to the nature of the study design, prospective double-blinding is impossible to maintain for Segment 2, Period B and Period C. However, effort shall be made to maintain a single blind (subjects blinded as to treatment assignment) during Period C.

At the Week 52/End of Study visit, all subjects remaining on treatment in Segment 2 will be offered the opportunity to enroll in a companion open-label long-term safety and efficacy trial of piclidenoson 3 mg BID for up to an additional 4 years.

Disease will be assessed using PASI, sPGA, the percentage of BSA involved, DLQI and PSSD, and, where applicable, PSSI and/or NAPSI.

Subjects enrolled in Segment 1 of the trial will return for efficacy and safety assessments and a new supply of study medication at Weeks 4 and 8; will be contacted remotely for safety monitoring at Weeks 2 and 12; and the final study assessments will be done at Week 16.

Subjects enrolled in Segment 2 of the trial will return for efficacy and safety assessments and a new supply of study medication at Weeks 4, 8, 16, 20, 24, 32, 36, 44; will be contacted remotely for safety monitoring at Weeks 2, 12, 28, 40, and 48; and will then have the final study assessments at Week 52.

PK assessment is applicable for the patients enrolled in Segment 2 only. Dose proportionality, effects of gender, age, renal function, and body weight on the PK parameters will be assessed if data permit. PK will be assessed through sparse sampling.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years and above;
2. Diagnosis of moderate-to-severe chronic plaque-type psoriasis with BSA involvement ≥10%;
3. PASI score ≥12 at the Screening and Baseline visits;
4. Static PGA ≥3 at the Screening and Baseline visits;
5. Candidate for systemic treatment or phototherapy for psoriasis;
6. Duration of psoriasis of at least 12 months;
7. Females of childbearing potential must have a negative serum pregnancy test at screening;
8. Female subjects of childbearing potential must use at least one acceptable contraceptive method throughout the course of the trial and for 1 month after the last dose of study medication;
9. Male subjects must refrain from sperm donation during treatment and until at least 1 month after the last dose of study medication. Male subjects must agree to use condoms throughout the course of the trial and for 1 month after the last dose of study medication;
10. Ability to complete the study in compliance with the protocol; and
11. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Psoriasis limited to erythrodermic, guttate, palmar, plantar, or generalized pustular psoriasis in the absence of plaque psoriasis;
2. Treatment with systemic retinoids, systemic corticosteroids, tofacitinib, apremilast, immunosuppressive agents (e.g., methotrexate, cyclosporine), or any other approved drugs for the indication of plaque psoriasis (e.g., deucravacitinib) within 4 weeks of the Baseline visit;
3. Treatment with a monoclonal antibody or other biologic agent for psoriasis within 8 weeks for etanercept, adalimumab, or infliximab, or within 12 weeks for all other agents, prior to the Baseline visit;
4. Treatment with Vitamin D analogs, keratolytics, coal tar (other than on the scalp, palms, groin, and/or soles), any topical corticosteroid, calcineurin inhibitors, vitamin A analogs, retinoids, anthralin, calcipotriene, tazarotene, methoxsalen, trimethyl-psoralens, fumarate, PDE4 inhibitors, or aryl hydrocarbon receptor-modulating agents within 2 weeks of the Baseline visit;
5. Ultraviolet or Dead Sea therapy within 4 weeks of the Baseline visit, or anticipated need for either of these therapies during the study period;
6. Treatment with lithium, hydroxychloroquine or chloroquine within 2 weeks of the Baseline visit, or anticipated need for such drugs during the study period, unless dose has been stable for 3 months prior to the Screening visit and will remain stable throughout the trial;
7. Estimated glomerular filtration rate (eGFR) ≥50 mL/min/1.73m2 by the Modification of Diet in Renal Disease equation at Screening (NOTE: In Segment 2, a renally-impaired subgroup of at least 10 12 subjects with eGFR of 20-49 mL/min/1.73m2 will be enrolled for PK analysis purposes);
8. Liver aminotransferase levels greater than 1.5 times the laboratory's upper limit of normal at Screening;
9. QTcF interval > 450 milliseconds (msec) for males or > 470 msec for females on Screening Visit and Baseline visit ECGs (average of triplicate ECGs at each visit) (except when QT prolongation is associated with right or left bundle branch block or cardiac pacemaker, in which case enrollment is allowed);
10. A condition which increases proarrhythmic risk, including hypokalemia, hypomagnesemia, or congenital Long QT Syndrome;
11. Ongoing or planned use of a concomitant medication that is on the CredibleMedsTM list of drugs known to cause Torsades des Pointes;
12. Active gastrointestinal disease which could interfere with the absorption of oral medication;
13. Pregnancy, planned pregnancy, lactation, or inadequate contraception as judged by the Investigator;
14. Active drug or alcohol dependence;
15. Concomitant use of strong cytochrome P450 inducers, e.g., rifampin, phenobarbital, phenytoin, carbamazepine;
16. PHQ-9 score ˃ 4 at baseline;
17. Any significant/uncontrolled neuropsychiatric illness judged as clinically significant by the investigator during screening or at Day 1, or any lifetime history of suicidal ideation, suicidal behavior, or suicidal attempts by medical history or by Columbia Suicide Severity Rating Scale (C-SSRS) documentation, or by answering "yes" to Question 4 or 5 for suicidal ideation on the C-SSRS at screening or at Day 1, or is clinically deemed to have a suicide risk by the investigator;
18. Previous participation in a piclidenoson (CF101) clinical trial;
19. Significant acute or chronic medical or psychiatric illness that, in the judgment of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study; and
20. Participation in another investigational drug or vaccine trial concurrently or within 30 days prior to the Screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects who achieve a Psoriasis Area and Severity Index (PASI) score response of ≥75% (PASI 75) | 16 weeks
  Improvement of psoriasis by 75% or more
proportion of subjects who achieve a Static Physician's Global Assessment (sPGA) of 0 or 1 with at least a 2-point improvement from Baseline | 16 weeks
  Improvement of psoriasis by physicians' judgment
Proportion of subjects who experience adverse events | 52 weeks
  All adverse events occurring the trial will be recorded

SECONDARY OUTCOMES:
Efficacy as determined by the proportion of subjects who achieve both PASI 75 and sPGA of 0 or 1 with at least a 2-point improvement from Baseline | 16 weeks
  Improvement of psoriasis by both assessment scales
Efficacy as determined by the proportion of subjects who achieve improvement of the Psoriasis Symptoms and Signs Diary (PSSD) to a score of 0 or 1 | 16 weeks
  Assessment of a quality of life measure
Efficacy as determined by the proportion of subjects who achieve improvement of the Dermatology Life Quality Index (DLQI) to a score of 0 or 1 | 16 weeks
  Assessment of a quality of life measure

IPD SHARING:
Plan to Share IPD: No